CLINICAL TRIAL: NCT02366962
Title: Phase III Study of ASP7374-Open-label Study of Subcutaneous Vaccination of Quadrivalent ASP7374 in Adult Subjects Aged 20 or Older
Brief Title: A Study to Assess the Safety of ASP7374 in Adult Subjects Aged 20 or Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UMN Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 7374-CL-0107
Record Dates: First submitted 2015-02-12; First posted 2015-02-19 (Estimated); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Influenza; Vaccine
Keywords: Influenza; Vaccine; ASP7374
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ASP7374 group (Experimental)
  Interventions: Biological: ASP7374

INTERVENTIONS:
Biological: ASP7374 — subcutaneous

SUMMARY:
The purpose of this study is to confirm the safety until Day 29 after injection of a single dose of quadrivalent vaccine ASP7374 in adult subjects aged 20 or older

ELIGIBILITY:
Inclusion Criteria:

* Medically stable, as judged on the basis of history and concurrent diseases
* Subject understands procedure of the protocol and is willing to comply with the protocol.

Exclusion Criteria:

* Scheduled to receive another vaccine during the study.
* Received influenza HA vaccine within 180 days prior to screening.
* Received or scheduled to receive a live vaccine within 28 days prior to vaccination with the study vaccine, and received or scheduled to receive an inactivated vaccine or a toxoid within 7 days prior to vaccination with the study vaccine.
* Diagnosis of immune deficit in the past has a family member (within the third degree of kinship) with a diagnosis of congenital immunodeficiency syndrome.
* Received one of the following medications or treatment prior to vaccination with the study vaccine:

  * 1. Within 28 days prior to vaccination with the study vaccine

    1. Interferon formulation
    2. Drugs which affect the immune system (e.g., immunosuppressants)
    3. Systemic corticosteroids and inhaled corticosteroids
    4. G-CSF and M-CSF
  * 2. Within 84 days prior to vaccination with the study vaccine

    1. Human immunoglobulin products
    2. Blood products
    3. Blood transfusion
  * 3. Within 180 days prior to vaccination with the study vaccine

    1. High-dose human immunoglobulin products (≥200 mg/kg)
* History of anaphylactic shock or an allergic reaction such as generalized eruption due to food or drug (including vaccines) allergies, fever ≥39.0°C within 2 days after the previous vaccination (influenza vaccine and others)
* History of seizures (exclude a pyrexial attack in childhood)
* History of Guillain-Barre syndrome or acute disseminated encephalomyelitis (ADEM)
* Body temperature of ≥37.5°C on Day 1 (before vaccination)
* Moderate to severe acute or febrile illness (≥37.5°C) within 7 days prior to vaccination
* Concurrent hepatic disease (exclude fatty liver, hepatic cyst, biliary stone and gallbladder poly, which have laboratory findings only, no clinical symptoms, and not necessary to treat), or AST (GOT) and/or ALT (GPT) of >100 IU/L at screening on Day 1
* Concurrent renal disease (exclude rental cyst and calculus kidney which have laboratory findings only, no clinical symptoms, and not necessary to treat), or creatinine of > 1.5 mg/dL at screening
* Concurrent respiratory disease, hematologic disease, or developmental disorders
* Concurrent or previous heart disease
* Concurrent or previous cerebrovascular disorder
* Concurrent malignancy or diagnosis or treatment of malignancy within 5 years before screening
* Diagnosis of mental disorder including schizophrenia, bipolar disorder, or major depressive disorder or cognitive impairment, or received medications for cognitive impairment
* Concurrent disease interfering with the evaluation of local and systemic reactions

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-02; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Safety assessed by adverse events | Up to Day 29

SECONDARY OUTCOMES:
Local and systemic reactions associated with the vaccination | Up to Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Fukuoka, Japan